CLINICAL TRIAL: NCT01979328
Title: The Efficacy of a Neuromuscular Stimulation Device (Geko™) in Promoting Blood Flow in a Plaster Cast as a Way of Offering Mechanical DVT Prophylaxis
Brief Title: Geko™ Plaster Cast Study, Deep Vein Thrombosis (DVT) Prophylaxis
Acronym: THRIVE-III
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: THRIVE-III
Record Dates: First submitted 2013-10-21; First posted 2013-11-08 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-10

CONDITIONS: Deep Vein Thrombosis
Keywords: Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — Casts, Surgical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study arm (Experimental): geko neuromuscular electrostimulation
  Interventions: Device: geko; Device: Plaster cast

INTERVENTIONS:
Device: geko
Device: Plaster cast

SUMMARY:
The primary objective of this study is to examine the flow characteristics of deep venous flow in the leg veins using Doppler ultrasound imaging and how this flow is modified by the application of a plaster and with a geko™ device in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Be in good general health and fitness.
2. Aged between 18 and 65 years.
3. Free of significant abnormal findings as determined by medical history (specifically an absence of DVT or haematological disorders or indications), screening physical examination, vital signs (sitting blood pressure, sitting pulse rate, sitting respiratory rate and body temperature) and duplex ultrasound)
4. BMI between 18 and 34
5. No history or signs of drug abuse (including alcohol), licit or illicit.
6. Has not used any medications (prescribed or over-the-counter including herbal remedies) judged to be significant by the Principal Investigator during the thirty (30) days preceding the study, and agrees not to use any medications during the course of the study without informing the Research Team.
7. Able to understand the Volunteer Information Sheet and signed the written Informed Consent Forms.
8. Able and willing to follow the Protocol requirements.

Exclusion Criteria:

1. Previous leg fracture. (within the last 12 months)
2. Any evidence of organ dysfunction, or any clinically significant deviation from normal in the physical determinations.
3. History or signs of haematological disorders (especially in relation to clotting or coagulation or previous Deep or superficial vein thrombosis/pulmonary embolism) or familiar history of such.
4. Peripheral arterial disease (ABPI<0.9), clinically significant varicose veins or lower limb ulceration.
5. Musculoskeletal disorders (such as pain during exercise of lower limb, rheumatoid or osteoarthritis).
6. Neurological disorders,(such as stroke, multiple sclerosis)
7. Recent surgery (such as abdominal, gynaecological, hip knee replacement).
8. Recent trauma to lower limbs.
9. Chronic Obesity (BMI Index >34).
10. Pregnancy.
11. Any Medication judged to be significant by the Principal Investigator.
12. Tobacco consumption
13. History of disorders of the gastrointestinal, hepatic, renal, cardiovascular, endocrine, neurological, dermatological, rheumatologic, metabolic (including diabetes), psychiatric, haematological (especially in relation to clotting or coagulation), or systemic disease judged to be significant.
14. A pulse rate of less than 50 beats/minute, a sitting systolic blood pressure >160 or <80 mmHg and/or a sitting diastolic pressure of >90 or <60 mmHg.
15. Any significant illness during the four (4) weeks preceding the screening period of the study.
16. Any contraindication to blood sampling.
17. Donation of blood during the eight (8) weeks preceding the screening period of the study or during the investigation.
18. Participation in any clinical study during the 8 weeks preceding the dosing period of the study
19. Fitted with a pacemaker or defibrillator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Blood flow | 4 hours

SECONDARY OUTCOMES:
microcirculatory blood flow | 4 hours

OTHER OUTCOMES:
acceptability and tolerance (composite endpoint) | 4 hours
  None validated questionnaire and a scoring index to assess comfort of the device

CONTACTS AND LOCATIONS:
Locations (1):
- Southampton University Hospital, Southampton, United Kingdom

REFERENCES:
- [Result] Warwick DJ, Shaikh A, Gadola S, Stokes M, Worsley P, Bain D, Tucker AT, Gadola SD. Neuromuscular electrostimulation viathe common peroneal nerve promotes lower limb blood flow in a below-kneecast: A potential for thromboprophylaxis. Bone Joint Res. 2013 Sep 2;2(9):179-85. doi: 10.1302/2046-3758.29.2000176. Print 2013. PMID 23999610